CLINICAL TRIAL: NCT01489189
Title: Prompt Panretinal Photocoagulation Versus Intravitreal Ranibizumab With Deferred Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Brief Title: Prompt Panretinal Photocoagulation Versus Ranibizumab+Deferred Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Acronym: Protocol S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRCR.net Protocol S
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-VEGF+Deferred PRP (Experimental): Anti-VEGF= Anti vascular endothelial growth factor. PRP= Panretinal photocoagulation. Intravitreal anti-VEGF with PRP only if indicated.
  Interventions: Drug: 0.5-mg Ranibizumab; Other: Deferred panretinal photocoagulation
- Prompt PRP (Active Comparator): PRP= Panretinal Photocoagulation. PRP alone.
  Interventions: Other: Prompt Panretinal Photocoagulation

INTERVENTIONS:
Other: Prompt Panretinal Photocoagulation — Panretinal photocoagulation alone at baseline (full session completed within 56 days).
  Arms: Prompt PRP
Drug: 0.5-mg Ranibizumab — Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline and up to every 4 weeks using defined retreatment criteria.
  Arms: Anti-VEGF+Deferred PRP
Other: Deferred panretinal photocoagulation — PRP is deferred until failure/futility criteria for intravitreal injection are met.
  Arms: Anti-VEGF+Deferred PRP

SUMMARY:
The primary objective of the protocol is to determine if visual acuity outcomes at 2 years in eyes with proliferative diabetic retinopathy (PDR) that receive anti-vascular endothelial growth factor (anti-VEGF) therapy with deferred panretinal photocoagulation (PRP) are non-inferior to those in eyes that receive standard prompt PRP therapy.

Secondary objectives include:

* Comparing other visual function outcomes (including Humphrey visual field testing and study participant self-reports of visual function) in eyes receiving anti-VEGF with deferred PRP with those in eyes receiving prompt PRP.
* Determining percent of eyes not requiring PRP when anti-VEGF is given in the absence of prompt PRP.
* Comparing safety outcomes between treatment groups.
* Comparing associated treatment and follow-up exam costs between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

Age >= 18 years -Individuals < 18 years old are not being included because proliferative diabetic retinopathy (PDR) is so rare in this age group that the diagnosis of PDR may be questionable.

Diagnosis of diabetes mellitus (type 1 or type 2)

Any one of the following will be considered to be sufficient evidence that diabetes is present:

* Current regular use of insulin for the treatment of diabetes
* Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
* Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria (see Procedures Manual for definitions) Able and willing to provide informed consent.

Meets at least all of the following ocular criteria criteria:

* Presence of PDR which the investigator intends to manage with PRP alone but for which PRP can be deferred for at least 4 weeks in the setting of intravitreal ranibizumab, in the investigator's judgment.
* Best corrected Electronic-Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity letter score > 24 (approximate Snellen equivalent 20/320) on the day of randomization.
* Media clarity, pupillary dilation, and study participant cooperation sufficient to administer PRP and obtain adequate fundus photographs and optical coherence tomography (OCT).

  * Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality

Exclusion Criteria:

Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.

A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).

* Individuals in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.

Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied.

* Study participants cannot receive another investigational drug while participating in the study.

Known allergy to any component of the study drug.

Blood pressure > 180/110 (systolic above 180 or diastolic above 110).

* If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.

Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.

Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.

* These drugs should not be used during the study.

For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.

* Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.

Individual is expecting to move out of the area of the clinical center to an area not covered by another Diabetic Retinopathy Clinical Research Network (DRCR.net) certified clinical center during the 3 years of the study.

Individual has any of the following ocular characteristics:

* History of prior panretinal photocoagulation (prior PRP is defined as ≥ 100 burns outside of the posterior pole)
* Tractional retinal detachment involving the macula.

  -- A tractional retinal detachment is not an exclusion if it is outside of the posterior pole (not threatening the macula) and in the investigator's judgment, is not a contraindication to intravitreal ranibizumab treatment and also does not preclude deferring PRP for at least 4 weeks in the setting of intravitreal ranibizumab
* Exam evidence of neovascularization of the angle (neovascularization of the iris alone is not an exclusion if it does not preclude deferring PRP for at least 4 weeks in the investigator's judgment).
* If macular edema is present, it is considered to be primarily due to a cause other than diabetic macular edema.

  -- An eye should not be considered eligible if:
  * macular edema is present that is considered to be related to ocular surgery such as cataract extraction or
  * clinical exam and/or OCT suggest that vitreoretinal interface abnormalities disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of any macular edema.
* An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).

  -- A vitreous or preretinal hemorrhage is not an exclusion if it is out of the visual axis and in the investigator's judgment is not having any affect on visual acuity.
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye were otherwise normal).
* History of intravitreal anti-VEGF treatment at any time in the past 2 months.
* History of corticosteroid treatment (intravitreal or peribulbar) at any time in the past 4 months.

  --If the investigator believes that there may still be a substantial effect 4 months after prior treatment (e.g., dose of intravitreal triamcinolone higher than 4 mg), the eye should not be included.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* History of (yttrium-aluminum-garnet) YAG capsulotomy performed within 2 months prior to randomization.
* Aphakia.
* Uncontrolled glaucoma (in investigator's judgment).
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Gross, MD, Study Chair — Carolina Retina Center
Locations (48):
- United States (48):
  - Retinal Consultants of AZ, Phoenix, Arizona
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - New England Retina Associates, Trumbull, Connecticut
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Ocala Eye Retina Consultants, Ocala, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Associates of Sarasota, Venice, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - North Shore University Health System, Glenview, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Retina Vitrous Center, Grand Blanc, Michigan
  - Barnes Retina Institute, St Louis, Missouri
  - Eye Surgical Associates, Lincoln, Nebraska
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - University of Rochester, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Family Eye Group, Lancaster, Pennsylvania
  - Retina Vitrous Consultants, Pittsburgh, Pennsylvania
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Spokane Eye Clinic, Spokane, Washington
  - Medical College of Wiconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Gross JG, Glassman AR. A Novel Treatment for Proliferative Diabetic Retinopathy: Anti-Vascular Endothelial Growth Factor Therapy. JAMA Ophthalmol. 2016 Jan;134(1):13-4. doi: 10.1001/jamaophthalmol.2015.5079. No abstract available. PMID 26583372
- [Background] Gross JG, Glassman AR. Panretinal Photocoagulation vs Anti-Vascular Endothelial Growth Factor for Proliferative Diabetic Retinopathy-Reply. JAMA Ophthalmol. 2016 Jun 1;134(6):716. doi: 10.1001/jamaophthalmol.2016.0703. No abstract available. PMID 27101313
- [Background] Beaulieu WT, Bressler NM, Melia M, Owsley C, Mein CE, Gross JG, Jampol LM, Glassman AR; Diabetic Retinopathy Clinical Research Network. Panretinal Photocoagulation Versus Ranibizumab for Proliferative Diabetic Retinopathy: Patient-Centered Outcomes From a Randomized Clinical Trial. Am J Ophthalmol. 2016 Oct;170:206-213. doi: 10.1016/j.ajo.2016.08.008. Epub 2016 Aug 12. PMID 27523491
- [Background] Bressler SB, Beaulieu WT, Glassman AR, Gross JG, Jampol LM, Melia M, Peters MA, Rauser ME; Diabetic Retinopathy Clinical Research Network. Factors Associated with Worsening Proliferative Diabetic Retinopathy in Eyes Treated with Panretinal Photocoagulation or Ranibizumab. Ophthalmology. 2017 Apr;124(4):431-439. doi: 10.1016/j.ophtha.2016.12.005. Epub 2017 Feb 1. PMID 28161147
- [Background] Hutton DW, Stein JD, Bressler NM, Jampol LM, Browning D, Glassman AR; Diabetic Retinopathy Clinical Research Network. Cost-effectiveness of Intravitreous Ranibizumab Compared With Panretinal Photocoagulation for Proliferative Diabetic Retinopathy: Secondary Analysis From a Diabetic Retinopathy Clinical Research Network Randomized Clinical Trial. JAMA Ophthalmol. 2017 Jun 1;135(6):576-584. doi: 10.1001/jamaophthalmol.2017.0837. PMID 28492920
- [Background] Gross JG, Glassman AR, Klein MJ, Jampol LM, Ferris FL 3rd, Bressler NM, Beck RW. Interim Safety Data Comparing Ranibizumab With Panretinal Photocoagulation Among Participants With Proliferative Diabetic Retinopathy. JAMA Ophthalmol. 2017 Jun 1;135(6):672-673. doi: 10.1001/jamaophthalmol.2017.0969. PMID 28492921
- [Background] Jampol LM, Odia I, Glassman AR, Baker CW, Bhorade AM, Han DP, Jaffe GJ, Melia M, Bressler NM, Tanna AP; Diabetic Retinopathy Clinical Research Network. PANRETINAL PHOTOCOAGULATION VERSUS RANIBIZUMAB FOR PROLIFERATIVE DIABETIC RETINOPATHY: Comparison of Peripapillary Retinal Nerve Fiber Layer Thickness in a Randomized Clinical Trial. Retina. 2019 Jan;39(1):69-78. doi: 10.1097/IAE.0000000000001909. PMID 29135802
- [Background] Bressler SB, Beaulieu WT, Glassman AR, Gross JG, Melia M, Chen E, Pavlica MR, Jampol LM; Diabetic Retinopathy Clinical Research Network. Panretinal Photocoagulation Versus Ranibizumab for Proliferative Diabetic Retinopathy: Factors Associated with Vision and Edema Outcomes. Ophthalmology. 2018 Nov;125(11):1776-1783. doi: 10.1016/j.ophtha.2018.04.039. Epub 2018 Jul 3. PMID 29980333
- [Background] Gross JG, Glassman AR, Liu D, Sun JK, Antoszyk AN, Baker CW, Bressler NM, Elman MJ, Ferris FL 3rd, Gardner TW, Jampol LM, Martin DF, Melia M, Stockdale CR, Beck RW; Diabetic Retinopathy Clinical Research Network. Five-Year Outcomes of Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA Ophthalmol. 2018 Oct 1;136(10):1138-1148. doi: 10.1001/jamaophthalmol.2018.3255. Erratum In: JAMA Ophthalmol. 2019 Apr 1;137(4):467. doi: 10.1001/jamaophthalmol.2019.0032. PMID 30043039
- [Background] Sun JK, Glassman AR, Beaulieu WT, Stockdale CR, Bressler NM, Flaxel C, Gross JG, Shami M, Jampol LM; Diabetic Retinopathy Clinical Research Network. Rationale and Application of the Protocol S Anti-Vascular Endothelial Growth Factor Algorithm for Proliferative Diabetic Retinopathy. Ophthalmology. 2019 Jan;126(1):87-95. doi: 10.1016/j.ophtha.2018.08.001. Epub 2018 Aug 7. PMID 30096354
- [Background] Bressler SB, Beaulieu WT, Glassman AR, Gross JG, Melia M, Chen E, Pavlica MR, Jampol LM; Diabetic Retinopathy Clinical Research Network. PHOTOCOAGULATION VERSUS RANIBIZUMAB FOR PROLIFERATIVE DIABETIC RETINOPATHY: Should Baseline Characteristics Affect Choice of Treatment? Retina. 2019 Sep;39(9):1646-1654. doi: 10.1097/IAE.0000000000002377. PMID 30807516
- [Background] Glassman AR, Beaulieu WT, Stockdale CR, Beck RW, Bressler NM, Labriola LT, Melia M, Oliver K, Sun JK. Effect of telephone calls from a centralized coordinating center on participant retention in a randomized clinical trial. Clin Trials. 2020 Apr;17(2):195-201. doi: 10.1177/1740774519894229. Epub 2020 Jan 27. PMID 31984762
- [Background] Maguire MG, Liu D, Glassman AR, Jampol LM, Johnson CA, Baker CW, Bressler NM, Gardner TW, Pieramici D, Stockdale CR, Sun JK; DRCR Retina Network. Visual Field Changes Over 5 Years in Patients Treated With Panretinal Photocoagulation or Ranibizumab for Proliferative Diabetic Retinopathy. JAMA Ophthalmol. 2020 Mar 1;138(3):285-293. doi: 10.1001/jamaophthalmol.2019.5939. PMID 31999300
- [Background] Hutton DW, Stein JD, Glassman AR, Bressler NM, Jampol LM, Sun JK; DRCR Retina Network. Five-Year Cost-effectiveness of Intravitreous Ranibizumab Therapy vs Panretinal Photocoagulation for Treating Proliferative Diabetic Retinopathy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2019 Dec 1;137(12):1424-1432. doi: 10.1001/jamaophthalmol.2019.4284. PMID 31647496
- [Result] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Derived] Talcott KE, Valentim CCS, Hill L, Stoilov I, Singh RP. Baseline Diabetic Retinopathy Severity and Time to Diabetic Macular Edema Resolution with Ranibizumab Treatment: A Meta-Analysis. Ophthalmol Retina. 2023 Jul;7(7):605-611. doi: 10.1016/j.oret.2023.02.003. Epub 2023 Feb 10. PMID 36774994
- [Derived] Maguire MG, Liu D, Bressler SB, Friedman SM, Melia M, Stockdale CR, Glassman AR, Sun JK; DRCR Retina Network. Lapses in Care Among Patients Assigned to Ranibizumab for Proliferative Diabetic Retinopathy: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Dec 1;139(12):1266-1273. doi: 10.1001/jamaophthalmol.2021.4103. PMID 34673898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with 2 eyes in the study had 1 eye randomly assigned to receive ranibizumab and 1 eye to receive panretinal photocoagulation.
  Two-year completed visits include those that occurred between 644 and 812 days (between 92 and 116 weeks).
Groups:
- Anti-VEGF+Deferred PRP: Anti vascular endothelial growth factor (Anti-VEGF). Panretinal photocoagulation (PRP). Intravitreal anti-VEGF with PRP only if indicated.
  0.5-mg Ranibizumab: Intravitreal injection of 0.5 mg ranibizumab (Lucentis™) at baseline and up to every 4 weeks using defined retreatment criteria.
  Deferred panretinal photocoagulation: PRP is deferred until failure/futility criteria for intravitreal injection are met.
- Prompt PRP: Panretinal Photocoagulation (PRP). PRP alone.
  Prompt Panretinal Photocoagulation: Panretinal photocoagulation alone at baseline (full session completed within 56 days).
Period: Overall Study
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Started | 191 (Number of Eyes) | 203 (Number of Eyes)
Completed | 160 (Number of Eyes) | 168 (Number of Eyes)
Not Completed | 31 | 35
Not completed — Withdrawal by Subject | 20 | 23
Not completed — Death | 10 | 8
Not completed — Missed Visit | 1 | 4

BASELINE CHARACTERISTICS:
Population: Units in Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP | Total
Number analyzed (Participants) | 191 | 203 | 394
Age, Customized [Median (Inter-Quartile Range); unit: years] | 52 [44 to 59] | 51 [44 to 59] | 51 [44 to 59]
Sex/Gender, Customized [Number; unit: eyes]
  Female | 83 | 92 | 175
  Male | 108 | 111 | 219
Race/Ethnicity, Customized [Number; unit: eyes]
  White | 100 | 101 | 201
  Hispanic | 48 | 51 | 99
  Black/African American | 38 | 43 | 81
  Asian | 2 | 3 | 5
  American Indian/Alaskan Native | 1 | 0 | 1
  More than 1 race | 0 | 2 | 2
  Unknown/not reported | 2 | 3 | 5
Number of study eyes [Number; unit: eyes]
  One | 102 | 114 | 216
  Two (one in each group) | 89 | 89 | 178
Diabetes Type [Number; unit: eyes]
  Type 1 | 43 | 41 | 84
  Type 2 | 140 | 155 | 295
  Uncertain | 8 | 7 | 15
Duration of Diabetes [Median (Inter-Quartile Range); unit: years] | 18 [12 to 24] | 17 [11 to 23] | 18 [11 to 24]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: percent] — Hemoglobin A1c data were missing for 7 in the anti-VEGF+Deferred PRP group and 5 in the prompt PRP group.
  percent | 8.6 [7.5 to 10.4] | 8.9 [7.5 to 10.4] | 8.7 [7.5 to 10.4]
Prior Myocardial Infarction [Number; unit: eyes] | 3 | 4 | 7
Prior Stroke [Number; unit: eyes] | 4 | 3 | 7
Arterial Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 99 [88 to 108] | 99 [88 to 107] | 99 [88 to 108]
Visual Acuity [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  letters | 75 (12.8) | 75.2 (12.5) | 75.1 (12.6)
Optical Coherence Tomography Central Subfield Thickness [Median (Inter-Quartile Range); unit: µm] — OCT central subfield thickness measurements were missing for 2 in the anti-VEGF+deferred PRP group and 2 in the prompt PRP group.
  Assessments from OCT machines other than Zeiss Stratus were converted to equivalent on Zeiss Stratus machines.
  µm | 223 [196 to 271] | 230 [203 to 265] | 229 [199 to 266]
Presence of Center-Involved Diabetic Macular Edema with Visual Acuity Impairment [Number; unit: eyes] — OCT central subfield thickness measurements were missing for 2 in the anti-VEGF+deferred PRP group and 2 in the Prompt PRP group.
  eyes | 42 | 46 | 88
Presence of Center-Involved Diabetic Macular Edema Regardless of Visual Acuity [Number; unit: eyes] — OCT central subfield thickness measurements were missing for 2 in the anti-VEGF+deferred PRP group and 2 in the Prompt PRP group.
  eyes | 55 | 62 | 117
Neovascularization on Clinical Examination [Number; unit: eyes]
  Of the disc | 96 | 103 | 199
  Elsewhere | 166 | 174 | 340
Phakic Lens Status on Clinical Exam [Number; unit: eyes] | 170 | 187 | 357
Diabetic Retinopathy Severity [Number; unit: eyes] — Diabetic retinopathy level data were missing for 2 in the anti-VEGF+deferred PRP group and 4 in the prompt PRP group. Proliferative diabetic retinopathy (PDR) could not be identified by the reading center in 46 eyes (12%) but was subsequently confirmed by other imaging modes in 29 (63%) of the 46 eyes.
  eyes
    Microaneurysms only (level 20) | 0 | 1 | 1
    Mild NPDR (level 35) | 6 | 4 | 10
    Moderate NPDR (level 43) | 2 | 5 | 7
    Moderately severe NPDR (level 47) | 10 | 15 | 25
    Severe NPDR (level 53) | 1 | 1 | 2
    Prior PRP without active PDR (level 60) | 0 | 1 | 1
    Mild PDR (level 61) | 30 | 31 | 61
    Moderate PDR (level 65) | 68 | 67 | 135
    High-risk PDR (levels 71 and 75) | 69 | 73 | 142
    Advanced PDR, macular center attached (level 81) | 2 | 0 | 2
    Advanced PDR, macular center detached (level 85) | 1 | 1 | 2
Prior treatment for diabetic macular edema (DME) [Number; unit: eyes] | 43 | 36 | 79
Prior focal/grid laser treatment for DME [Number; unit: eyes] | 30 | 29 | 59
Prior anti-VEGF treatment for DME [Number; unit: eyes] | 21 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity From Baseline
Description: Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart.
Time Frame: 2-years
Population: Participants that completed the 2-year visit.
Measure: Mean (95% Confidence Interval); unit: letters
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 160 | 168
Number analyzed (Eyes) | 160 | 168
letters | 2.8 [0.4 to 5.2] | 0.2 [-1.9 to 2.3]

2. Secondary Outcome: Mean Visual Acuity
Description: as for outcome 1
Time Frame: 2-years
Population: Participants that completed the 2-year visit.
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 160 | 168
Number analyzed (Eyes) | 160 | 168
letters | 78.7 (16.3) | 76.2 (14.1)

3. Secondary Outcome: Number of Eyes With Greater Than or Equal to 10 Letter Vision Gain
Time Frame: 2-years
Population: Eyes with a baseline letter score of 78 or less (approximate Snellen equivalent 20/32 or worse) from participants that completed the 2-year visit.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 81 | 86
Number analyzed (Eyes) | 81 | 86
eyes | 35 | 31

4. Secondary Outcome: Humphrey Visual Field Test Cumulative Score Change From Baseline
Description: Visual fields, collected using the Humphrey Visual Field analyzer, measured the total point score (sum of retinal sensitivities of all points) tested on 30-2 and 60-4 patterns, which included the mid-peripheral and peripheral visual fields. A lower score indicates greater visual field loss.The cumulative score is the sum of all visual field sensitivity values for each of the four individual quadrants of the visual field (the quadrants are divided by the horizontal and vertical lines). The range can be from 0 to about 600 for the 30-2 test [for each quadrant], and from 0 to about 400 or 450 for the peripheral test.
Time Frame: 2-years
Population: Humphrey visual fields were obtained at a subset of sites. Fields with excessive false positive response, excessive false negative response, or excessive fixation loss were excluded from analysis. Twenty-two eyes in the anti-VEGF+deferred PRP group and 25 eyes in the prompt PRP group were excluded.
Measure: Median (Inter-Quartile Range); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 58 | 57
Number analyzed (Eyes) | 58 | 57
decibels | -25 [-232 to 223] | -379 [-723 to -75]

5. Secondary Outcome: Frequency of Vitrectomy
Time Frame: 2-years
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 191 | 203
Number analyzed (Eyes) | 191 | 203
eyes | 8 | 30

6. Secondary Outcome: Mean Change in OCT Central Subfield Thickness From Baseline
Description: All baseline and 2-year optical coherence tomography (OCT) scans were evaluated by the OCT reading center.
Time Frame: 2-years
Population: Eyes with optical coherence tomography (OCT) data at baseline and 2-years.
Measure: Mean (95% Confidence Interval); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 149 | 161
Number analyzed (Eyes) | 149 | 161
µm | -47 [-61 to -33] | -3 [-15 to 9]

7. Secondary Outcome: Development of Central DME With Vision Impairment by 2-years
Time Frame: 2-years
Population: Excludes that did not have central DME with vision impairment (20/32 or worse) at baseline.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 147 | 155
Number analyzed (Eyes) | 147 | 155
eyes | 15 | 42

8. Secondary Outcome: Number of Eyes With Vitreous Hemorrhage
Time Frame: 2-years
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 191 | 203
Number analyzed (Eyes) | 191 | 203
Eyes | 52 | 69

9. Secondary Outcome: Number of Eyes Without Active or Regressed Neovascularization on Fundus Photography at 2-years
Time Frame: 2-years
Population: Eyes with baseline diabetic retinopathy level 61B or worse (active neovascularization). Last-observation-carried-forward was used for 23 eyes in the anti-VEGF+Deferred PRP group and 25 eyes in the Prompt PRP group missing photographs at 2 years if 1-year fundus photographs were available.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 142 | 148
Number analyzed (Eyes) | 142 | 148
eyes | 49 | 44

10. Secondary Outcome: Number of Eyes With Greater Than or Equal to 10 Letter Vision Loss
Time Frame: 2-year
Population: Participants that completed the 2-year visit.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Anti-VEGF+Deferred PRP | Prompt PRP
Number analyzed (Participants) | 160 | 168
Number analyzed (Eyes) | 160 | 168
eyes | 15 | 23

ADVERSE EVENTS:
Groups:
- Bilateral Participants: Participants with one eye enrolled in each arm of the study.
Arm/Group | Bilateral Participants | Anti-VEGF+Deferred PRP | Prompt PRP
Serious Adverse Events (participants affected / at risk) | 36/89 | 50/102 | 43/114
Other Adverse Events (participants affected / at risk) | 85/89 | 96/102 | 105/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bilateral Participants (N=89) | Anti-VEGF+Deferred PRP (N=102) | Prompt PRP (N=114)
Leukaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 6 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1 | 1
Coronary artery restenosis (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 3 | 2
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Diabetes mellitus (Endocrine disorders) | 0 | 2 | 0
Diabetes mellitus inadequate control (Endocrine disorders) | 1 | 2 | 1
Diabetic ketoacidosis (Endocrine disorders) | 0 | 4 | 3
Hyperglycaemia (Endocrine disorders) | 2 | 0 | 0
Hypoglycaemia (Endocrine disorders) | 1 | 1 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Endophthalmitis (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastroenteritis viral (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest pain (General disorders) | 2 | 5 | 3
Death (General disorders) | 1 | 3 | 2
Hernia (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Abscess (Infections and infestations) | 1 | 1 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 1 | 1
Localised infection (Infections and infestations) | 4 | 3 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine abnormal (Investigations) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Fractured coccyx (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Brain neoplasm (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 3 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Vertigo (Nervous system disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 0 | 1
Pyelonephritis (Renal and urinary disorders) | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 7 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 4 | 3
Renal impairment (Renal and urinary disorders) | 0 | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Gangrene (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cardiac operation (Surgical and medical procedures) | 1 | 0 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 1
Knee operation (Surgical and medical procedures) | 0 | 0 | 2
Leg amputation (Surgical and medical procedures) | 0 | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 1 | 1
Surgery (Surgical and medical procedures) | 1 | 1 | 0
Toe amputation (Surgical and medical procedures) | 0 | 3 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Carotid artery disease (Vascular disorders) | 0 | 0 | 1
Cerebrovascular accident (Vascular disorders) | 1 | 2 | 3
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3
Hypotension (Vascular disorders) | 1 | 1 | 0
Ischaemic stroke (Vascular disorders) | 0 | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Transient ischaemic attack (Vascular disorders) | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than .00001% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bilateral Participants (N=89) | Anti-VEGF+Deferred PRP (N=102) | Prompt PRP (N=114)
Anaemia (Blood and lymphatic system disorders) | 7 | 9 | 6
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphoedema (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 5 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1
Ear infection (Ear and labyrinth disorders) | 1 | 4 | 2
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1 | 0
Otitis media acute (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0
Diabetes mellitus (Endocrine disorders) | 3 | 3 | 2
Diabetes mellitus inadequate control (Endocrine disorders) | 7 | 5 | 4
Diabetic ketoacidosis (Endocrine disorders) | 0 | 0 | 1
Hyperglycaemia (Endocrine disorders) | 3 | 6 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypoglycaemia (Endocrine disorders) | 1 | 8 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 0
Thyroid neoplasm (Endocrine disorders) | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 1
Accommodation disorder (Eye disorders) | 1 | 0 | 0
Altered visual depth perception (Eye disorders) | 0 | 0 | 2
Angle closure glaucoma (Eye disorders) | 2 | 0 | 0
Anterior chamber cell (Eye disorders) | 3 | 1 | 1
Anterior chamber flare (Eye disorders) | 0 | 0 | 2
Aphakia (Eye disorders) | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 0 | 1
Blepharal papilloma (Eye disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 3 | 2 | 0
Blepharospasm (Eye disorders) | 0 | 2 | 0
Cataract (Eye disorders) | 8 | 15 | 17
Cataract cortical (Eye disorders) | 3 | 3 | 4
Cataract nuclear (Eye disorders) | 0 | 5 | 6
Cataract subcapsular (Eye disorders) | 7 | 8 | 5
Chalazion (Eye disorders) | 0 | 2 | 1
Chemical eye injury (Eye disorders) | 0 | 1 | 0
Chorioretinal disorder (Eye disorders) | 0 | 1 | 1
Choroidal detachment (Eye disorders) | 0 | 0 | 1
Choroiditis (Eye disorders) | 2 | 0 | 0
Colour blindness acquired (Eye disorders) | 0 | 1 | 0
Conjunctival cyst (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 10 | 16 | 9
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 2 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1
Conjunctivitis viral (Eye disorders) | 0 | 0 | 1
Corneal abrasion (Eye disorders) | 3 | 1 | 2
Corneal defect (Eye disorders) | 1 | 0 | 1
Corneal disorder (Eye disorders) | 0 | 1 | 0
Corneal epithelium defect (Eye disorders) | 1 | 0 | 0
Corneal erosion (Eye disorders) | 1 | 1 | 0
Corneal oedema (Eye disorders) | 2 | 2 | 5
Corneal pigmentation (Eye disorders) | 0 | 1 | 0
Corneal scar (Eye disorders) | 1 | 0 | 0
Cystoid macular oedema (Eye disorders) | 1 | 2 | 2
Diabetic retinal oedema (Eye disorders) | 9 | 6 | 8
Diabetic retinopathy (Eye disorders) | 0 | 4 | 5
Diplopia (Eye disorders) | 5 | 2 | 0
Dry eye (Eye disorders) | 12 | 10 | 8
Episcleritis (Eye disorders) | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 3 | 0
Eye infection (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 8 | 9 | 3
Eye pain (Eye disorders) | 22 | 14 | 21
Eye penetration (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 7 | 8 | 11
Eye swelling (Eye disorders) | 1 | 1 | 0
Eyelid disorder (Eye disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 3 | 3 | 3
Eyelid ptosis (Eye disorders) | 1 | 2 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 1 | 4
Giant papillary conjunctivitis (Eye disorders) | 1 | 0 | 0
Glare (Eye disorders) | 1 | 4 | 0
Glaucoma (Eye disorders) | 7 | 4 | 3
Halo vision (Eye disorders) | 0 | 0 | 1
Hyphaema (Eye disorders) | 3 | 2 | 1
Hypotony of eye (Eye disorders) | 0 | 1 | 0
Iris adhesions (Eye disorders) | 1 | 1 | 0
Iris neovascularisation (Eye disorders) | 3 | 3 | 2
Iritis (Eye disorders) | 1 | 0 | 3
Keratitis (Eye disorders) | 0 | 1 | 0
Keratopathy (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 6 | 3 | 9
Lenticular pigmentation (Eye disorders) | 1 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 1 | 0
Macular fibrosis (Eye disorders) | 13 | 10 | 9
Macular hole (Eye disorders) | 0 | 0 | 2
Macular ischaemia (Eye disorders) | 5 | 0 | 1
Macular oedema (Eye disorders) | 2 | 5 | 7
Metamorphopsia (Eye disorders) | 5 | 1 | 0
Ocular discomfort (Eye disorders) | 2 | 4 | 4
Ocular hyperaemia (Eye disorders) | 4 | 1 | 7
Ocular hypertension (Eye disorders) | 2 | 1 | 3
Optic atrophy (Eye disorders) | 0 | 0 | 1
Optic nerve cupping (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 7 | 5 | 3
Photopsia (Eye disorders) | 10 | 7 | 5
Posterior capsule opacification (Eye disorders) | 1 | 4 | 2
Punctate keratitis (Eye disorders) | 2 | 2 | 4
Pupillary block (Eye disorders) | 0 | 1 | 0
Pupillary reflex impaired (Eye disorders) | 0 | 0 | 1
Retinal aneurysm (Eye disorders) | 2 | 1 | 0
Retinal artery embolism (Eye disorders) | 0 | 2 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 12 | 13 | 19
Retinal disorder (Eye disorders) | 1 | 2 | 0
Retinal exudates (Eye disorders) | 4 | 8 | 0
Retinal haemorrhage (Eye disorders) | 10 | 12 | 8
Retinal ischaemia (Eye disorders) | 0 | 2 | 2
Retinal neovascularisation (Eye disorders) | 9 | 15 | 14
Retinal oedema (Eye disorders) | 1 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1
Retinal vascular disorder (Eye disorders) | 1 | 2 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 1 | 0
Scleritis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 33 | 25 | 26
Visual acuity reduced (Eye disorders) | 17 | 20 | 20
Visual field defect (Eye disorders) | 1 | 1 | 2
Visual impairment (Eye disorders) | 9 | 8 | 4
Vitreal cells (Eye disorders) | 1 | 1 | 0
Vitreous adhesions (Eye disorders) | 3 | 3 | 0
Vitreous detachment (Eye disorders) | 6 | 4 | 9
Vitreous disorder (Eye disorders) | 2 | 1 | 0
Vitreous floaters (Eye disorders) | 38 | 32 | 35
Vitreous haemorrhage (Eye disorders) | 37 | 46 | 49
Vitreous opacities (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colon cancer (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastroenteritis viral (Gastrointestinal disorders) | 3 | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 6 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Lactose intolerance (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 9 | 6
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tooth abscess (Gastrointestinal disorders) | 2 | 1 | 0
Tooth infection (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5 | 2
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 3 | 3 | 2
Chills (General disorders) | 0 | 1 | 1
Device related infection (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 1
Flank pain (General disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1
Injection site irritation (General disorders) | 0 | 1 | 1
Local swelling (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 5 | 4 | 6
Pain (General disorders) | 1 | 2 | 3
Pyrexia (General disorders) | 1 | 2 | 0
Swelling (General disorders) | 2 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 5 | 4 | 5
Abscess (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 2 | 0
Gingival infection (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 3 | 2
Influenza (Infections and infestations) | 7 | 11 | 7
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 5 | 0
Onychomycosis (Infections and infestations) | 2 | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 1 | 0
Biopsy skin (Investigations) | 0 | 1 | 0
Blood creatinine abnormal (Investigations) | 0 | 1 | 0
Blood glucose decreased (Investigations) | 2 | 0 | 1
Blood glucose increased (Investigations) | 2 | 0 | 0
Blood testosterone decreased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 6 | 4 | 4
Laboratory test abnormal (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 4 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 1 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot fracture (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Gout (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Hand fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Meniscus injury (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Multiple fractures (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Concussion (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 3 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 5 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 15 | 10 | 18
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1 | 0
IVth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 2 | 1
Nerve injury (Nervous system disorders) | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Temporal arteritis (Nervous system disorders) | 0 | 1 | 0
Vertigo (Nervous system disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 3
Depression (Psychiatric disorders) | 2 | 1 | 8
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Stress (Psychiatric disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 2 | 0
Bladder cancer (Renal and urinary disorders) | 1 | 0 | 0
Cystitis (Renal and urinary disorders) | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Kidney infection (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Pyelonephritis (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 5 | 2 | 3
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 3 | 0 | 5
Renal impairment (Renal and urinary disorders) | 1 | 1 | 1
Renal osteodystrophy (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 4 | 6 | 4
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Prostate cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine leiomyoma (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 15 | 17 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 7
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 3 | 4 | 1
Contusion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Excoriation (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Onychomycosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin papilloma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Menopause (Social circumstances) | 0 | 0 | 1
Abdominal panniculectomy (Surgical and medical procedures) | 0 | 1 | 0
Benign tumour excision (Surgical and medical procedures) | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 4 | 2
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 0 | 0 | 1
Gastric banding (Surgical and medical procedures) | 0 | 0 | 1
Glaucoma surgery (Surgical and medical procedures) | 1 | 0 | 0
Retinal laser coagulation (Surgical and medical procedures) | 1 | 3 | 1
Skin lesion excision (Surgical and medical procedures) | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 3 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 3 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 6 | 8
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 13 | 24 | 18
Hypotension (Vascular disorders) | 2 | 1 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
Transient ischaemic attack (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results can not be discussed until they have been made available to the public.